CLINICAL TRIAL: NCT00732810
Title: A Randomized Phase 2 Study of SCH 727965 in Subjects With Advanced Breast and Non Small Cell Lung (NSCLC) Cancers
Brief Title: SCH 727965 in Patients With Advanced Breast and Lung Cancers (Study P04716)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04716
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Breast Neoplasms; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — dinaciclib; Capecitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Breast cancer randomized to SCH 727965 (Experimental)
  Interventions: Drug: SCH 727965
- Breast cancer randomized to capecitabine (Active Comparator)
  Interventions: Drug: Capecitabine
- SCH 727965 in breast cancer after progression on capecitabine (Experimental)
  Interventions: Drug: SCH 727965
- NSCLC randomized to SCH 727965 (Experimental): Note: Enrollment of participants with NSCLC was completed per protocol as of 26 JAN 2010
  Interventions: Drug: SCH 727965
- NSCLC randomized to erlotinib (Active Comparator): Note: Enrollment of participants with NSCLC was completed per protocol as of 26 JAN 2010
  Interventions: Drug: Erlotinib
- SCH 727965 in NSCLC after progression on erlotinib (Experimental): Note: Crossover to SCH 727965 after progression on erlotinib was completed per protocol as of 26 JAN 2010
  Interventions: Drug: SCH 727965

INTERVENTIONS:
Drug: SCH 727965 — SCH 727965 50 mg/m^2 IV on Day 1 of each 21 day cycle until disease progression.
  Arms: Breast cancer randomized to SCH 727965; NSCLC randomized to SCH 727965; SCH 727965 in NSCLC after progression on erlotinib; SCH 727965 in breast cancer after progression on capecitabine
Drug: Capecitabine — Capecitabine 1250 mg/m^2 orally twice daily from Day 1 to Day 14 of each 21 day cycle until disease progression.
  Other Names: Xeloda
  Arms: Breast cancer randomized to capecitabine
Drug: Erlotinib — Erlotinib 150 mg orally once daily until disease progression.
  Other Names: Tarceva
  Arms: NSCLC randomized to erlotinib

SUMMARY:
To determine the activity of SCH 727965 in participants with breast cancer and in participants with nonsmall-cell lung cancer (NSCLC) compared to standard treatment. The standard treatment used is capecitabine for breast cancer and erlotinib for NSCLC. The study will also determine the activity of SCH 727965 treatment in participants who experience cancer progression after standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years, either sex, any race.
* Histologically or cytologically confirmed breast cancer or NSCLC; and radiographic or clinically advanced disease.
* BREAST CANCER:

  * participant must have previously received both a taxane and an anthracycline (unless anthracycline therapy is contraindicated) in the adjuvant and/or metastatic setting,
  * participant with HER2-positive disease must have progressed after trastuzumab and concomitant or subsequent lapatinib,
  * participant must have received at least one, but no more than two prior regimens for recurrent or metastatic disease (endocrine and biologic therapies do not count as chemotherapeutic regimens).
* NSCLC: at least one, but no more than two prior chemotherapeutic regimens for advanced disease.
* Measurable disease by the RECIST.
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
* Adequate hematologic, renal, and hepatic organ function and laboratory parameters.
* Ability to swallow tablets.

Exclusion Criteria:

* Known brain metastases. For NSCLC only, a participant with central nervous system metastasis is eligible provided the participant has received definitive local therapy (ie, radiation therapy or surgery), has stopped receiving treatment with corticosteroids, and is without symptoms for at least 4 weeks before randomization.
* History of previous radiation therapy to >25% of total bone marrow.
* Known HIV infection.
* Known active hepatitis B or hepatitis C.
* Previous treatment with SCH 727965 or other cyclin-dependent-kinase inhibitors.
* BREAST CANCER:

  * known dihydropyrimidine dehydrogenase deficiency,
  * previous treatment with capecitabine.
* NSCLC: previous treatment with erlotinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Time to disease progression. | Every 6 weeks for 30 weeks, and then every 9 weeks. Assessments continue until disease progression.
  Date of randomization to date of tumor progression.
Overall response rate in participants treated with SCH 727965 after disease progression on the comparator drug. | Every 6 weeks for 30 weeks, and then every 9 weeks.
  Percentage of participants with tumor responses (partial responses + complete responses).

REFERENCES:
- [Result] Mita MM, Joy AA, Mita A, Sankhala K, Jou YM, Zhang D, Statkevich P, Zhu Y, Yao SL, Small K, Bannerji R, Shapiro CL. Randomized phase II trial of the cyclin-dependent kinase inhibitor dinaciclib (MK-7965) versus capecitabine in patients with advanced breast cancer. Clin Breast Cancer. 2014 Jun;14(3):169-76. doi: 10.1016/j.clbc.2013.10.016. Epub 2013 Oct 26. PMID 24393852
- [Result] Stephenson JJ, Nemunaitis J, Joy AA, Martin JC, Jou YM, Zhang D, Statkevich P, Yao SL, Zhu Y, Zhou H, Small K, Bannerji R, Edelman MJ. Randomized phase 2 study of the cyclin-dependent kinase inhibitor dinaciclib (MK-7965) versus erlotinib in patients with non-small cell lung cancer. Lung Cancer. 2014 Feb;83(2):219-23. doi: 10.1016/j.lungcan.2013.11.020. Epub 2013 Dec 2. PMID 24388167